CLINICAL TRIAL: NCT01171651
Title: A Phase 2 Open-Label Pilot Safety Study of JX-594 (Vaccinia GM-CSF/Thymidine Kinase-Deactivated Virus) Administered by IV Infusion Followed by Intratumoral Injection Prior to Standard Sorafenib Treatment in Patients With Unresectable Primary Hepatocellular Carcinoma
Brief Title: A Study of Recombinant Vaccinia Virus Prior to Sorafenib to Treat Unresectable Primary Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jennerex Biotherapeutics (Industry)
Responsible Party: Sponsor
Organization: SillaJen, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JX594-HEP016
Record Dates: First submitted 2010-07-26; First posted 2010-07-28 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2011-06

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Vaccinia; Vaccinia Virus; JX-594; Jennerex; Primary Hepatocellular Carcinoma; Primary Liver Cancer; Liver Cancer; Sorafenib; Nexavar; Pexa-Vec
MeSH Terms: conditions — Carcinoma, Hepatocellular; Vaccinia; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- JX-594 followed by sorafenib (Experimental): 1e9 pfu (plaque-forming units) total JX-594 dose on each of up to four (4) JX-594 treatment days. Sorafenib is initiated after 3 JX-594 treatments and briefly interrupted if an optional 4th JX-594 treatment is given.
  Interventions: Drug: JX-594 followed by sorafenib

INTERVENTIONS:
Drug: JX-594 followed by sorafenib — Patients will receive a total dose of 1e9 per treatment starting with one IV dose on Day 1 and injected intratumorally in 1-5 intrahepatic tumors on Day 8 and 22. Starting on Day 25 (3 days after the final JX-594 dose) patients will initiate oral sorafenib therapy twice daily according to standard approved guidelines. An optional maintenance JX-594 dose may be given intratumorally at Week 12 (sorafenib briefly interrupted).

SUMMARY:
The purpose of this pilot safety study is to evaluate the safety and tolerability of JX-594 (Pexa-Vec) administered intravenously and intratumorally prior to standard sorafenib therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation or clinical/laboratory diagnosis of primary hepatocellular carcinoma (HCC)
* Cancer is not surgically resectable for cure
* Child Pugh A or B
* Performance Score: KPS score of ≥ 70
* Platelet count ≥ 50,000 plts/mm3
* Total bilirubin ≤ 2.5 x ULN
* AST, ALT < 5.0 x ULN
* Acceptable coagulation status: INR ≤ 1.5 x ULN
* Acceptable kidney function: Serum creatinine < 2.0 mg/dL
* Sorafenib naive or refractory to sorafenib therapy Tumor Status: At least one intrahepatic tumor, and at least ≥50% of the total intrahepatic viable tumor mass, measurable by CT and injectable under imaging-guidance (note: injected and/or viable tumors must be previously untreated or ≥20% increase in size since preceding local-regional treatment).

Exclusion Criteria:

* Known contraindications to sorafenib
* Pregnant or nursing an infant
* Significant immunodeficiency due to underlying illness (e.g. hematological malignancies, congenital immunodeficiencies and/or HIV infection/AIDS) and/or medication (e.g. high-dose systemic corticosteroids)
* History of exfoliative skin condition (e.g. severe eczema, ectopic dermatitis, or similar skin disorder) that at some stage has required systemic therapy
* Clinically significant and/or rapidly accumulating ascites, peri-cardial and/or pleural effusions
* Severe or unstable cardiac disease
* Current, known CNS malignancy
* Use of anti-platelet or anti-coagulation medication
* Use of the following anti-viral agents: ribavirin, adefovir, cidofovir (within 7 days prior to the first treatment), and PEG-IFN (within 14 days prior to the first treatment).
* Patients with household contacts who meet any of these criteria unless alternate living arrangements can be made during the patient's active dosing period and for 7 days following the last dose of study medication:
* Pregnant or nursing an infant
* Children < 12 months old
* History of exfoliative skin condition that at some stage has required systemic therapy
* Significant immunodeficiency due to underlying illness (e.g. HIV/AIDS) and/or medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-08; Primary Completion 2013-02 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Determine safety and tolerability of intravenous infusion of JX-594 followed by intratumoral injections with JX-594 prior to standard sorafenib therapy | Safety evaluations through 28 days after last dose of JX-594
  Adverse events will be collected and assessed to assess safety and tolerability through 28 days after last dose of JX-594 (or until all events considered probably or possibly related to JX-594 have resolved, stabilized, or returned to baseline status).

SECONDARY OUTCOMES:
Determine Disease Control Rate (DCR) at 12 weeks | Disease control and response assessment at 12 weeks from first JX-594 dose
  DCR: confirmed complete response, partial response or stable disease based on modified RECIST and/or Choi response criteria
Determine radiographic response rate | Periodically throughout study participation (average of up to 1 year)
  Response rate evaluation based on modified RECIST and/or Choi response criteria
Determine overall survival time | Ongoing (average of 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: David H Kirn, MD, Study Director — Jennerex Biotherapeutics
Locations (2):
- South Korea (2):
  - Pusan National University Hospital, Busan
  - Pusan National University Yangsan Hospital, Yangsan

REFERENCES:
- [Derived] Breitbach CJ, Arulanandam R, De Silva N, Thorne SH, Patt R, Daneshmand M, Moon A, Ilkow C, Burke J, Hwang TH, Heo J, Cho M, Chen H, Angarita FA, Addison C, McCart JA, Bell JC, Kirn DH. Oncolytic vaccinia virus disrupts tumor-associated vasculature in humans. Cancer Res. 2013 Feb 15;73(4):1265-75. doi: 10.1158/0008-5472.CAN-12-2687. Epub 2013 Feb 7. PMID 23393196
- See also: Sponsor Company Website — http://www.jennerex.com